CLINICAL TRIAL: NCT06623916
Title: Can Elastographic Evaluation Be a New Approach in Prediction of Endometrial Cancer Prognostic Markers?
Brief Title: Strain-elastography in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Alper seyhan (Other)
Responsible Party: Sponsor-Investigator, Alper seyhan, assoc. prof., Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Other Study IDs: 2022-179
Record Dates: First submitted 2024-09-23; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Endometrial Cancer
Keywords: elastography; endometrial cancer; prognosis
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Endometrial Cancer Survivors — strain sonoelastograghy method has not been studied before in endometrial cancer as a prognostic factor. we compared well known pathologic prognostic factors with elastographic methods.

SUMMARY:
Strain elastography is a novel, non-invasive, easy applicable method to determine the tissue characteristics of benign or malign lesions in various organs. In this preliminary prospective study, we investigated the relation between the known pathological prognostic factors of endometrial cancer and elastographic characteristics of tumor tissue

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic cancer, particularly in developed countries of the World. Today, it ranks as the 4th most common cancer among the women after breast, colorectal and lung malignencies. Although 4% of patients are premenopausal, most common symptom of disease is postmenopausal bleeding. Obtaining pathological sample as an endometrial Pipelle Biopsy, dilatation-curettage or hysterescopic excision are main diagnostic methods in endometrial cancer. Prognosis of disease depends on age, grade, myometrial invasion-histologic type of tumor, lymph node and distant metastasis.

In addition to pathologic reports; transvaginal ultrasound is most commonly used preoperative non invasive, no radiation-related and low cost imaging method to assess the endometrial cavity, endo-myometrial invasion, tumor diameter, cervical and adnexal involvement. Some of these risk factors can be easily detected with transvaginal ultrasound as well as intraoperative frozen-section examination.

Sonoelastography is a novel technique, which evaluate tissue stiffness both qualitatively and quantitatively and can distinguish different lesions in various organs as liver, breast and thyroid. Strain and shear-wave imagings are two main elastographic technics that commonly used with ultrasound technology. In the first method, the operator exerts manual compression on the tissue with the ultrasound transducer. Strain elastography evaluates the tissue elasticity by measuring the degree of distorsion by the compression and decompression of soft tissues and strain ratio (SR) is obtained by proportioning the tissue elasticity of the suspicious pathologic area with a reference point. Manual compression works fairly well for superficial organs such as the breast, superficial lymph nodes and thyroid but is challenging for assessing elasticity in deeper located organs such as the liver. Strain elastography is a semi-quantitative method due to the variations in compression and decompression pressures and selected ROI areas between practitioners. The use of SR makes this relative subjective technic more objective. In shear wave elastography, the ultrasound transducer is held steady, and tissue displacement is generated by internal physiologic motion (e.g. cardiovascular, respiratory). Since this method is not dependent on superficially applied compression, variations between practitioners are negligible and it may be used to assess deeper located organs.

In gynecology clinical practice, sono elastography has been used in recent years in different subjects as ovarian and endometrial benign lesions. In diagnostic process, elastography is not been well established in endometrial cancer.

In this study, we aimed to determine whether sonoelastography could be a new prognostic predictor in endometrial cancer. Accordingly, we examined the relationship between the elastographic features of the lesions and known pathologic prognostic factors in endometrial cancer cases.

Inform consent was provided from all patients before evaluation. Biopsy-confirmed ( Pipelle sampling or dilatation and curettage ) 90 endometrial cancer patients were evaluated. Diagnosis of different types of tumors in the last 5 years, presence of synchronous malignancy, presence of non epithelial uterine tumor, lack of patient data, presence of full-thickness uterine and cervical involvement (lack of evaluation for elastography), lack of patient compliance for transvaginal ultrasound and inoperable cases (lack of definitive pathologic report) were the exclusion criterias of the study. Demographic and clinical datas were collected through a questionnaire including age, gravida, parity, weight (kg), height (cm). Body mass index (BMI)was calculated as a kg/ cm2. Cancer Antigen-125(CA-125) values were recorded as a IU/ml. Positron emission tomography/computed tomography (PET/CT) imaging was performed before surgery for evaluating of distant metastasis and excluding inoperable patients. Standardized Uptake Values (SUV)-max value of tumor in uterus was recorded. 63 patients who met the criteria were evaluated with transvaginal ultrasound and strain elastography mode of ultrasound. Before the measurements, strain elastography technique was defined and figures were added to ensure reproducibility. The strain measurements are displayed as a semitransparent color map called an elastogram, which is overlaid on the b-mode image. Typically, low strain (stiff tissue) is displayed in blue, and high strain (soft tissue) is displayed in red, although the color scale can vary depending on the ultrasound vendor. A pseudo-quantitative measurement called the strain ratio can be used, which is the ratio of strain measured in adjacent (usually normal) reference tissue region of interest (ROI) to strain measured in a target lesion ROI. SR >1 indicates that the target lesion compresses less than the normal reference tissue, indicating lower strain and greater stiffness. With these general information, cervix and uterus were examined in sagittal plane in all patients with transvaginal b-mode ultrasonography and elastography mode on the day before surgery. The size of the lesion in the cavity, the degree of myometrial invasion, possible presence of cervical and adnexal involvement were evaluated. The reason why the uterine cervix and intact myometrium were chosen as reference points is that they are adjacent to the target lesion and can be evaluated in the same window in elastography mode. After the elastography window was opened, the reference (intact myometrial area and cervical area) and target (endometrial lesion) ROI were determined, compression and decompressions cycles were applied with the transvaginal probe in one-second periods to create a pressure tracing. Strain ratio was calculated at the peak of the pressure in the area where the trace was regular. Comparison between intact myometrium and target tissue was defined as 'strain-corpus', while comparison between cervix and target tissue was defined as 'strain ratio-cervix'. Strain ratios were calculated at least 3 times and mean strain ratio was saved. All ultrasound examinations were performed by a single gynecologist oncologist and Voluson S8 (GE Healthcare, Wisconsin, USA) equipped with a 4.0-9.0 MHz multifrequency transvaginal probe was used for examination. When the definitive pathology results of the cases were reported in the postoperative period; tumor diameter, grade, myoinvasion, cervical involvement, lymph node metastasis and distant metastasis datas were recorded. According to the prognostic factors specified in pathology report, endometrial cancer risk groups defined by ESGO-ESMO-ESTRO guidelines were determined as a low- intermediate - high risk.

Datas were analyzed using SPSS 21.0 (SPSS, Chicago, IL, USA) statistical program. The distribution of continuous variables was analyzed with using visual and analytic method (Kolmogorov-Smirnov/Shapiro-Wilk test). Mean and standart deviations were used in normal distribution, while median and min-max values were used in non-normal distribution. Chi-square test was used to show the difference between categorical variables. Pearson and Spearman's rank correlation analyzes were used for continuous variables. Student-t Test and Kruskal Wallis analysis was used to compare the continuous variables in independent groups. The receiver operating characteristics (ROC) analysis was used to determine whether the mean strain ratio values had a statistically significant effect on the differentiation in prognostic factors. p < 0.05 was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epitheliel endometrial cancer diagnosis with biopsy.

Exclusion Criteria:

* Diagnosis of different types of tumors in the last 5 years
* Presence of synchronous malignancy, presence of non epithelial uterine tumor
* Lack of patient data
* Presence of full-thickness uterine and cervical involvement (lack of evaluation for elastography)
* Lack of patient compliance for transvaginal ultrasound
* Inoperable cases (lack of definitive pathologic report)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with endometrial cancer diagnosis will be operated in gynaecologic oncology clinic in Adnan Menderes University
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
feasibility; to compare the stiffness and strain character of tumor tissue with well-known pathological prognostic factors of endometrial cancer. | strain ratio measurements of tumor tissue were performed one night before the operation. these data were compared with pathological reports which results 1 month after the cytoreductive surgery.
  The strain measurements are displayed as a semitransparent color map called an elastogram, which is overlaid on the b-mode image. Typically, low strain (stiff tissue) is displayed in blue, and high strain (soft tissue) is displayed in red, although the color scale can vary depending on the ultrasound vendor. A pseudo-quantitative measurement called the strain ratio can be used, which is the ratio of strain measured in adjacent (usually normal) reference tissue region of interest (ROI) to strain measured in a target lesion ROI. SR &gt;1 indicates that the target lesion compresses less than the normal reference tissue, indicating lower strain and greater stiffness.The receiver operating characteristics (ROC) analysis was used to determine whether the mean strain ratio values had a statistically significant effect on the differentiation in well known pathological prognostic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Department of Gynaecologic Oncology, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data available on request due to privacy/ethical restrictions

REFERENCES:
- [Background] Ong CL, Chew LE, Han NR, Ooi CC, Yeo YC, Chew SH, Wong WL, Tang PH, Teo SY. The Characteristics of Real-time Transvaginal Sono-elastography in Endometrial Cancer. J Med Ultrasound. 2022 Jan 6;30(2):101-108. doi: 10.4103/JMU.JMU_74_21. eCollection 2022 Apr-Jun. PMID 35832355